CLINICAL TRIAL: NCT02352688
Title: A Randomised Controlled Trial on Preoperative Elderly Patients Undergoing Colorectal Cancer Surgery With Enhanced Geriatric Input
Brief Title: RCT on Elderly Patients Undergoing Colorectal Cancer Surgery With Enhanced Geriatric Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tony Wing Chung Mak, Assistant Professor in Colorectal Surgery, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2014.550-T
Record Dates: First submitted 2015-01-19; First posted 2015-02-02 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Colorectal Cancer
Keywords: elderly; enhanced recovery after surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Colorectal Geriatric Care (Active Comparator): Multidisciplinary team involving in the elderly colorectal cancer patients' pre-, peri- and postoperative care.
  Interventions: Procedure: Enhanced Colorectal Geriatric Care
- Standard Surgical Care (No Intervention): Standard care given to elderly patients undergoing colorectal cancer resection.

INTERVENTIONS:
Procedure: Enhanced Colorectal Geriatric Care
  Arms: Enhanced Colorectal Geriatric Care

SUMMARY:
This study evaluates the effects of enhanced geriatric input on elderly patients undergoing colorectal cancer surgery. Half of the participants will received additional pre, peri and post-operative care from the geriatric team, while the other half will receive standard surgical care.

DETAILED DESCRIPTION:
Additional geriatric care involves appropriate assessments and interventions by a multidisciplinary team involving geriatricians, physiotherapist, occupational therapist, surgical team, dietician and social worker. It is divided into three stages of care: 1) preoperative assessment, 2) perioperative care and 3) discharge or rehabilitation. In preoperative assessment, a comprehensive geriatric assessment will be carried out which encompasses patients medical and social backgrounds, cognitive status, nutritional assessment and risk factors identification. Perioperative care includes a joint care by surgical and geriatric teams aiming to prevent and treat any postoperative complications. Discharge and rehabilitation aim to identifies and facilities any potential discharge problem or accelerates patients for rehabilitation to the appropriate locations.

Standard surgical care will be given to patients who are undergoing colorectal cancer surgery but without the additional input mentioned above.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive colorectal cancer patients (aged 70 and over) undergoing elective colorectal cancer surgery at the Prince of Wales Hospital, Shatin, Hong Kong
2. American Society of Anaesthesiologists fitness score of I, II or III

Exclusion Criteria:

1. Colorectal cancer patients aged 69 or under undergoing colorectal surgery
2. Patients undergoing emergency colorectal cancer resection
3. Patients with benign pathology
4. Patients with evidence of locally advanced or metastatic spread of their primary disease
5. Patient who are unable to give informed consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-05; Primary Completion 2017-05 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Length of postoperative hospital stay | up to 90 days

SECONDARY OUTCOMES:
30-day morbidity | 30 day from time of surgery
30-day mortality | 30 day from time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tony Mak, MD, Principal Investigator — Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong SAR, China
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong